CLINICAL TRIAL: NCT03817892
Title: Assessment of the Impact of Relay Timing and CPRmeter Guidance on the Quality of External Chest Compression: Compression Is Life In Cardiac Arrest - Human Study (CILICA-HS).
Brief Title: Compression Is Life In Cardiac Arrest - Human Study (CILICA-HS).
Acronym: CILICA-HS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2018-A02000-55; 17-248 (Other: CHU Caen)
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation
Keywords: No-Flow; Chest Compression Fraction; Out Hospital; External Chest Compression Relay; External Chest Compression Guidance; External Chest Compression Quality; Correct Compression Score
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: This is a randomized, multicenter, open-label study using a 2x2 factorial design comparing (i) the rhythm of External Chest Compression relays every 4 minutes versus every 2 minutes on the Chest Compression Fraction; (ii) the use of real-time guidance of the External Chest Compression via a feedback device (CPRmeter®) versus no guidance on the quality of the External Chest Compression (correct compression score).
Masking Description: The participants being in cardiac arrest at the time of the performance of the study, they are not aware of the arm of randomization in which they are initialy and they are inform as soon as their clinical status allow it.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unguided 2 minutes (U2) (No Intervention): The External Chest Compression are performed without guidance of the CPRmeter device (according to the current guidelines).
  The duration or rhythm of a relay during which a rescuer performs External Chest Compression before being relayed by another rescuer is 2 minutes according to the current guidelines.
- Unguided 4 minutes (U4) (Experimental): The External Chest Compression are performed without guidance of the CPRmeter device (according to the current guidelines).
  The duration or rhythm of a relay during which a rescuer performs External Chest Compression before being relayed by another rescuer is 4 minutes. (Rhythm of a relay 4 minutes)
  Interventions: Other: Rhythm of a relay 4 minutes
- Guided 2 minutes (G2) (Experimental): The External Chest Compression are performed with guidance of the CPRmeter device. (Guidance of the External Chest Compression) The duration or rhythm of a relay during which a rescuer performs External Chest Compression before being relayed by another rescuer is 2 minutes according to the current guidelines.
  Interventions: Other: Guidance of the External Chest Compression
- Guided 4 minutes (G4) (Experimental): The External Chest Compression are performed with guidance of the CPRmeter device. (Guidance of the External Chest Compression) The duration or rhythm of a relay during which a rescuer performs External Chest Compression before being relayed by another rescuer is 4 minutes. (Rhythm of a relay 4 minutes)
  Interventions: Other: Guidance of the External Chest Compression; Other: Rhythm of a relay 4 minutes

INTERVENTIONS:
Other: Guidance of the External Chest Compression — The CPRmeter® device is positioned on the patient's chest with a disposable adhesive. In the situation of guidance of the External Chest Compression the rescuers have access in real time on the screen to visual feedback on the quality of the External Chest Compression performed and indications of possible corrections to improve the quality of the External Chest Compression . In the case of non-guidance of the External Chest Compression , a mask is position on the screen in order to hide the feedback information.
  Other Names: CPRmeter's feedback
  Arms: Guided 2 minutes (G2); Guided 4 minutes (G4)
Other: Rhythm of a relay 4 minutes — The duration or rhythm of a relay is the time during which a rescuer performs External Chest Compression before being relayed by another rescuer. This time is 2 minutes in non intervention group according to the current guidelines and 4 minutes in experimental group.
  Arms: Guided 4 minutes (G4); Unguided 4 minutes (U4)

SUMMARY:
The management of out-of-hospital cardiac arrest is complex and multifactorial. With an incidence between 5 and 15 per 10,000 (46,000 patients per year in France) and a survival rate of only 5% to 15%, the room for improvement remains significant even today and is based on fast and optimal care. Thus French and international recommendations insist on the central element of external chest compression (ECC) and especially its quality (Monsieurs KG and Al. Resuscitation 2015; 95: 1-80). Improving the chest compression fraction (CCF) by limiting time without cardiac massage (No-Flow) is a second major point of the recommendations (Vaillancourt C and Al. Resuscitation 2011; 82: 1501-7). The survival of cardiac arrest victims is closely related on this No-Flow time. The principle of the chain of survival (early warning - ECC - defibrillation - resuscitation) implies that the deterioration of a single link threaten the whole of the care. To meet these qualitative needs, ECC guidance devices have been developed. They make possible to improve the quality of the ECC achieved (Hostler D and Al. BMJ 2011; 342d512). Their use is one of the areas of improvement mentioned in the recommendations. Our team studied in simulation the prolonged effects of guidance on the quality of the ECC during a prolonged resuscitation, with encouraging results (Buléon C and Al. Am J Emerg Med 2016; 34: 1754-60). The investigators propose a study evaluating the efficiency of the guidance of the ECC and the impact of the time of relay on the CCF. The investigators formulate two hypotheses that they wish to test simultaneously using a 2x2 factorial design, in a multicenter randomized trial. The first assumption is that a 4-minute relay rate improves the CCF (by reducing the No-Flow time) compared to the currently recommended 2-minute relay rate. The second hypothesis is that a guiding device improves the quality of the ECC.

This study should, over a period of 2 years, include 500 patients with cardiac arrest for whom specialized resuscitation is undertaken. The investigators hope by this study to improve the knowledge on the optimal rhythm of the ECC and to validate "in vivo" the interest for the guidance found on manikin. This study should make it possible to clarify the recommendations with a high level of evidence in this field and thus contribute to improving the prognosis of the victims of an out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
The management of out-of-hospital cardiac arrest is complex and multifactorial. With an incidence between 5 and 15 per 10,000 (46,000 patients per year in France) and a survival rate of only 5% to 15%, the room for improvement remains significant even today and is based on fast and optimal care. Thus French and international recommendations insist on the central element of external chest compression (ECC) and especially its quality (Monsieurs KG and Al. Resuscitation 2015; 95: 1-80). Improving the chest compression fraction (CCF) by limiting time without cardiac massage (No-Flow) is a second major point of the recommendations (Vaillancourt C and Al. Resuscitation 2011; 82: 1501-7). The survival of cardiac arrest victims is closely related on this No-Flow time. The principle of the chain of survival (early warning - ECC - defibrillation - resuscitation) implies that the deterioration of a single link threaten the whole of the care. To meet these qualitative needs, ECC guidance devices have been developed. They make possible to improve the quality of the ECC achieved (Hostler D and Al. BMJ 2011; 342d512). Their use is one of the areas of improvement mentioned in the recommendations. Our team studied in simulation the prolonged effects of guidance on the quality of the ECC during a prolonged resuscitation, with encouraging results (Buléon C and Al. Am J Emerg Med 2016; 34: 1754-60). The investigators propose a study evaluating the efficiency of the guidance of the ECC and the impact of the time of relay on the CCF. The investigators formulate two hypotheses that they wish to test simultaneously using a 2x2 factorial design, in a multicenter randomized trial. The first assumption is that a 4-minute relay rate improves the CCF (by reducing the No-Flow time) compared to the currently recommended 2-minute relay rate. The second hypothesis is that a guiding device improves the quality of the ECC.

This study should, over a period of 2 years, include 500 patients with cardiac arrest for whom specialized resuscitation is undertaken. The investigators hope by this study to improve the knowledge on the optimal rhythm of the ECC and to validate "in vivo" the interest for the guidance found on manikin. This study should make it possible to clarify the recommendations with a high level of evidence in this field and thus contribute to improving the prognosis of the victims of an out-of-hospital cardiac arrest.

Cardiac arrest (CA) remains a challenge for pre-hospital care. With an incidence of between 5 and 15 per 10,000 (46,000 patients per year in France) and a survival rate of only 5% to 15%, there is yet room for improvement in treatment to reduce morbi-mortality of these patients. The quality of cardiopulmonary resuscitation (CPR) is at the heart of the last three five-year recommendations. (1-3) The latest recommendations emphasize the importance for professionals to work at the highest quality of CPR and External Chest Compression (ECC) possible. (3) The ratio of the time during which the ECC is performed (Low-Flow) to the total time of the resuscitation is referred to as the Chest Compression Fraction (CCF). During CPR, it is essential for the patient's survival to minimize ECC disruption times and therefore to increase the CCF, as this is an independent element in CA survival's improvement. (4,5) ECC interruptions are deleterious to at least two titles. First, they are a source of direct stop in cerebral and coronary perfusions potentially altering the neurological prognosis and the probability of Return of Spontaneous Circulation. (6) Secondly, the quality of the cardiac output generated by the ECC at the time of resuming of the ECC after an interruption is less good for more than 30 seconds: time need for that several chest compressions can restore the best flow possible. (6,7) Reducing these interruptions and improving the ECC is therefore a major goal of improving CPR. The guidelines are that CCF must be greater than 60% and some experts estimate that a CCF of 80% is possible. (8,9) The outcome of patients with pre-hospital CA is significantly, positively and independently correlated with the consistency to different CCF targets, ECC frequency, ECC depth, and brief pre-external electric shock pause (<10 seconds). (10) There is evidence that ECC's guidance improves adequacy to guidelines and allows to be closer with the ECC frequency, depth and release objectives. (11) The investigators have proved in simulation that the guidance of the ECC delays the deterioration of the overall quality of the ECC and its components (frequency, depth and relaxation) related to fatigue during a prolonged ECC beyond the 2 ECC relay minutes currently recommended. (12) Strategies to get closer with the guidelines regarding the quality of the ECC associated with an improvement in CCF should add or even enhance their beneficial effects for the management of CA victims. Achieving high quality CPR requires the measurement of quality of CPR (ECC and CCF). (13,14) This idea of a support strategy enhanced by "bundles" of concepts is developing in the literature. Thus Cheskes S et al. Describe a "high quality CPR" such as the association of a CCF greater than 70% and achievement of the objectives of the recommendations for the frequency and depth of the ECC. (15) The place of devices for guiding the quality of the ECC needs to be specified. Indeed, studies of their use in real-life situations are criticized for their methodological qualities and their size. (16) The use of a real-time guidance device is proposed as a possibility in the latest guidelines without being an indispensable element due to the lack of current evidence. (3) Its use or non-use does not imply any obvious loss of chance for patients. Evidence as to its usefulness therefore remains to be sought.

For this reason, the investigators wish, through an original, randomized, multi-center study, to provide some answers to the questions about the possibility of an improvement in CCF by the lengthening of the time between two ECC relays and the effect of guidance on the quality of the ECC. The design of the study will also allow to approach a possible combined effect of ECC relays rhythm and guidance. The currently recommended duration of a two-minute ECC cycle between two relays does not have a consistent evidence based and corresponds to a duration for which the ECC effort can be maintained in principle with efficiency. (3) Objective measures have shown that the quality of the ECC can be maintained beyond 2 minutes. Extending the duration of an ECC cycle could reduce the number of ECC interruptions and thus improve the CCF.

The investigators therefore formulate two hypotheses that they wish to test simultaneously using a 2x2 factorial design, in a multicenter randomized trial. The first assumption is that a 4-minutes relay rhythm improves the CCF (by reducing the No-Flow time) compared to the currently recommended 2-minutes relay rhythm. The second hypothesis is that a guiding device improves the quality of the ECC.

The CPRmeter® (guidance device used in this study) will record data on the ECC and its quality (depth, frequency, relaxation, CPRmeter® use time, No-Flow time and Low-Flow time) as well as ECC guidance for the group which will benefit from it (the other group will have the screen masked by a screen cap).

This study should, over a period of 2 years, include 500 major patients presenting a non-traumatic CA for whom a specialized CPR is undertaken. The investigators hope by this study to improve the knowledge on the optimal rhythm of the CEE and to validate "in vivo" the interest for the guidance found on manikin. This study should clarify the guidelines with a high level of evidence in this area and thus contribute to improving the prognosis of victims of out-hospital CA.

ELIGIBILITY:
Inclusion Criteria:

* Major person
* Victim of a cardiorespiratory arrest
* Eligible for inclusion procedure in immediate life emergency
* Affiliated to the social security system

Exclusion Criteria:

* Minor person.
* Pregnant woman over 6 months old or breastfeeding.
* Known incurable disease.
* Palliative care in progress.
* Decision not to resuscitate from the patient (anticipated directives) or from the medical team.
* Traumatic cardiac arrest.
* Impossibility or contraindication to the use of the External Chest Compression guidance system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Chest Compression Fraction | 1 day
  The Chest Compression Fraction (in percentage) corresponds to the resuscitation time during which a External Chest Compression is performed (Low Flow) related to the patient's management time by the prehospital rescue team.
Correct Compression Score | 1 day
  The correct compression score (in percentage) corresponds to a External Chest Compression for which simultaneously the depth is correct (50 to 60 mm), the frequency is correct (100 to 120 / min) and the relaxation is correct (<2500 g) .

SECONDARY OUTCOMES:
Depth of External Chest Compression | 1 day
  The depth of External Chest Compression (in millimeters) continuously recorded by the guidance system (average and percentage correct).
Frequency of External Chest Compression | 1 day
  The frequency of External Chest Compression (in number of compression per minute) recorded continuously by the guidance system (average and percentage correct)....
Relaxation of External Chest Compression | 1 day
  The relaxation of External Chest Compression corresponds to the residual force (in grams) recorded continuously by the guidance system (average and percentage correct)
Subjective rescuers' fatigue | 1 day
  The subjective fatigue assessed by rescuers who performed External Chest Compression using the Borg scale (average of the Borg Scale values of rescuers)
The delays and durations of care | 1 day
  The delays and durations of care (in minutes and seconds) based on the following events: cardiac arrest time, start time of the External Chest Compression, start time of resuscitation by the prehospital rescue team, end time of resuscitation (ROSC or death of the patient).
No-Flow and Low-Flow times | 1 day
  The times (in minutes and seconds) of No-Flow (time during which no External Chest Compression is performed) and Low-Flow (time during which External Chest Compression is performed, generating a minimum flow rate of organs).
Recuperation of Spontaneous Circulation | 1 day
  The rate of Recuperation of Spontaneous Circulation (percentage).
survival at hospital arrival | 1 day
  The rate of survival at hospital arrival
Neuron Specific Enolase | Day 1 and day 3
  The serum Neuron Specific Enolase level (ng/mL)
Survival | Day 2 and one month.
  The survival rate.
Cerebral Performance Category Score | up to one month.
  Cerebral Performance Category Score as discribe in Wijdicks EFM et al. Neurology 2006;67:203-10.

OTHER OUTCOMES:
Demographic data | Day 1
  Demographic data of the population (sexe, age, suspect cause of cardiac arrest, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Clément BULEON, MD, Principal Investigator — University Hospital of Caen; Pierre-Yves GUEUGNIAUD, MD, PhD, Study Chair — University Hospital of Lyon; Eric ROUPIE, MD, PhD, Study Chair — University Hospital of Caen
Locations (11):
- France (11):
  - University Hospital of Caen, Caen, Normandy
  - University Hospital of Amiens, Amiens
  - Hospital of Cherbourg - Louis Pasteur, Cherbourg
  - Hospital of Elbeuf Louviers Val de Reuil, Elbeuf
  - Hospital Eure-Seine Evreux, Évreux
  - Hospital of Le Havre -, Le Havre
  - University Hospital of Lille, Lille
  - Hospital of Lisieux - Robert Bisson, Lisieux
  - University Hospital of Lyon, Lyon
  - University Hospital of Rouen, Rouen
  - Hospital of Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] International Liaison Committee on Resuscitation. 2005 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Part 4: Advanced life support. Resuscitation. 2005 Nov-Dec;67(2-3):213-47. doi: 10.1016/j.resuscitation.2005.09.018. No abstract available. PMID 16324990
- [Background] Nolan JP, Soar J, Zideman DA, Biarent D, Bossaert LL, Deakin C, Koster RW, Wyllie J, Bottiger B; ERC Guidelines Writing Group. European Resuscitation Council Guidelines for Resuscitation 2010 Section 1. Executive summary. Resuscitation. 2010 Oct;81(10):1219-76. doi: 10.1016/j.resuscitation.2010.08.021. No abstract available. PMID 20956052
- [Background] Monsieurs KG, Nolan JP, Bossaert LL, Greif R, Maconochie IK, Nikolaou NI, Perkins GD, Soar J, Truhlar A, Wyllie J, Zideman DA; ERC Guidelines 2015 Writing Group. European Resuscitation Council Guidelines for Resuscitation 2015: Section 1. Executive summary. Resuscitation. 2015 Oct;95:1-80. doi: 10.1016/j.resuscitation.2015.07.038. Epub 2015 Oct 15. No abstract available. PMID 26477410
- [Background] Christenson J, Andrusiek D, Everson-Stewart S, Kudenchuk P, Hostler D, Powell J, Callaway CW, Bishop D, Vaillancourt C, Davis D, Aufderheide TP, Idris A, Stouffer JA, Stiell I, Berg R; Resuscitation Outcomes Consortium Investigators. Chest compression fraction determines survival in patients with out-of-hospital ventricular fibrillation. Circulation. 2009 Sep 29;120(13):1241-7. doi: 10.1161/CIRCULATIONAHA.109.852202. Epub 2009 Sep 14. PMID 19752324
- [Background] Wik L, Olsen JA, Persse D, Sterz F, Lozano M Jr, Brouwer MA, Westfall M, Souders CM, Travis DT, Herken UR, Lerner EB. Why do some studies find that CPR fraction is not a predictor of survival? Resuscitation. 2016 Jul;104:59-62. doi: 10.1016/j.resuscitation.2016.04.013. Epub 2016 May 4. PMID 27155547
- [Background] Berg RA, Sanders AB, Kern KB, Hilwig RW, Heidenreich JW, Porter ME, Ewy GA. Adverse hemodynamic effects of interrupting chest compressions for rescue breathing during cardiopulmonary resuscitation for ventricular fibrillation cardiac arrest. Circulation. 2001 Nov 13;104(20):2465-70. doi: 10.1161/hc4501.098926. PMID 11705826
- [Background] Cunningham LM, Mattu A, O'Connor RE, Brady WJ. Cardiopulmonary resuscitation for cardiac arrest: the importance of uninterrupted chest compressions in cardiac arrest resuscitation. Am J Emerg Med. 2012 Oct;30(8):1630-8. doi: 10.1016/j.ajem.2012.02.015. Epub 2012 May 23. PMID 22633716
- [Background] Kleinman ME, Brennan EE, Goldberger ZD, Swor RA, Terry M, Bobrow BJ, Gazmuri RJ, Travers AH, Rea T. Part 5: Adult Basic Life Support and Cardiopulmonary Resuscitation Quality: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S414-35. doi: 10.1161/CIR.0000000000000259. No abstract available. PMID 26472993
- [Background] Perkins GD, Jacobs IG, Nadkarni VM, Berg RA, Bhanji F, Biarent D, Bossaert LL, Brett SJ, Chamberlain D, de Caen AR, Deakin CD, Finn JC, Grasner JT, Hazinski MF, Iwami T, Koster RW, Lim SH, Ma MH, McNally BF, Morley PT, Morrison LJ, Monsieurs KG, Montgomery W, Nichol G, Okada K, Ong ME, Travers AH, Nolan JP; Utstein Collaborators. Cardiac Arrest and Cardiopulmonary Resuscitation Outcome Reports: Update of the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest: A Statement for Healthcare Professionals From a Task Force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia); and the American Heart Association Emergency Cardiovascular Care Committee and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Resuscitation. 2015 Nov;96:328-40. doi: 10.1016/j.resuscitation.2014.11.002. Epub 2014 Nov 11. PMID 25438254
- [Background] Cheskes S, Schmicker RH, Rea T, Morrison LJ, Grunau B, Drennan IR, Leroux B, Vaillancourt C, Schmidt TA, Koller AC, Kudenchuk P, Aufderheide TP, Herren H, Flickinger KH, Charleston M, Straight R, Christenson J; ROC investigators. The association between AHA CPR quality guideline compliance and clinical outcomes from out-of-hospital cardiac arrest. Resuscitation. 2017 Jul;116:39-45. doi: 10.1016/j.resuscitation.2017.05.003. Epub 2017 May 2. PMID 28476474
- [Background] Hostler D, Everson-Stewart S, Rea TD, Stiell IG, Callaway CW, Kudenchuk PJ, Sears GK, Emerson SS, Nichol G; Resuscitation Outcomes Consortium Investigators. Effect of real-time feedback during cardiopulmonary resuscitation outside hospital: prospective, cluster-randomised trial. BMJ. 2011 Feb 4;342:d512. doi: 10.1136/bmj.d512. PMID 21296838
- [Background] Buleon C, Delaunay J, Parienti JJ, Halbout L, Arrot X, Gerard JL, Hanouz JL. Impact of a feedback device on chest compression quality during extended manikin CPR: a randomized crossover study. Am J Emerg Med. 2016 Sep;34(9):1754-60. doi: 10.1016/j.ajem.2016.05.077. Epub 2016 May 28. PMID 27349359
- [Background] Goodloe JM, Idris AH. Metrics save lives: value and hurdles faced. Curr Opin Crit Care. 2017 Jun;23(3):204-208. doi: 10.1097/MCC.0000000000000408. PMID 28379867
- [Background] Lin S, Scales DC. Cardiopulmonary resuscitation quality and beyond: the need to improve real-time feedback and physiologic monitoring. Crit Care. 2016 Jun 28;20(1):182. doi: 10.1186/s13054-016-1371-9. PMID 27349642
- [Background] Cheskes S, Byers A, Zhan C, Verbeek PR, Ko D, Drennan IR, Buick JE, Brooks SC, Lin S, Taher A, Morrison LJ; Rescu Epistry Investigators. CPR quality during out-of-hospital cardiac arrest transport. Resuscitation. 2017 May;114:34-39. doi: 10.1016/j.resuscitation.2017.02.016. Epub 2017 Feb 24. PMID 28242210
- [Background] Wallace SK, Abella BS, Becker LB. Quantifying the effect of cardiopulmonary resuscitation quality on cardiac arrest outcome: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2013 Mar 1;6(2):148-56. doi: 10.1161/CIRCOUTCOMES.111.000041. Epub 2013 Mar 12. PMID 23481533
- [Derived] Buleon C, Parienti JJ, Morilland-Lecoq E, Halbout L, Cesareo E, Dubien PY, Jardel B, Boyer C, Husson K, Andriamirado F, Benet X, Morel-Marechal E, Aubrion A, Muntean C, Dupire E, Roupie E, Hubert H, Vilhelm C, Gueugniaud PY; CILICA-HS study group. Impacts of chest compression cycle length and real-time feedback with a CPRmeter(R) on chest compression quality in out-of-hospital cardiac arrest: study protocol for a multicenter randomized controlled factorial plan trial. Trials. 2020 Jul 8;21(1):627. doi: 10.1186/s13063-020-04536-3. PMID 32641090